CLINICAL TRIAL: NCT03449186
Title: Interleukin-17 and Th17 Inducing Cytokines Exacerbate Periodontal Disease During Pregnancy and Postpartum
Brief Title: Th17 Inducing Cytokines Pregnancy and After Postpartum
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Veli Özgen Öztürk, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: BAP-2015
Record Dates: First submitted 2018-01-26; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy
Keywords: periodontitis; postpartum
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancy group: Women, who were in their second trimester (weeks 16-24) or third trimester (weeks 25-34)selected for the study. Saliva and GCF samples were collected and clinical periodontal measurements were made gently
  Interventions: Other: Saliva collection; Other: GCF collection
- Postpartum group: Postpartum women 6 months after giving birth recalled. Saliva and GCF samples were collected and clinical periodontal measurements were made.
  Interventions: Other: Saliva collection; Other: GCF collection

INTERVENTIONS:
Other: Saliva collection
Other: GCF collection

SUMMARY:
The aim of this study was to investigate salivary and gingival crevicular fluid (GCF) levels of IL-17A, IL-17E, IL-6 AND IL-23 during 2/3 trimester of pregnancy and after delivery.

DETAILED DESCRIPTION:
IL-17 have a synergytic effect with IL-6 and IL-23. IL-17A levels elevated with periodontal diseases. Many systemical chronic conditions such as atherosclerosis and cardiovascular disease, pregnancy may contribute increasing of IL-17 family cytokine.

ELIGIBILITY:
Inclusion Criteria:

* women 2 and 3 trimester of their pregnancy

Exclusion Criteria:

* any known systemic disease,
* periodontal treatment within the last six months,
* patients having less than 10 teeth,
* smokers,
* individuals with a BMI > 30 kg/m2,
* gestational diabetes and preeclampsia during pregnancy.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy women in second and third trimester
Study Population: All participants had 20 teeth present at least.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changing Il-17A levels | 6 month
  Salivary and GCF level measured by ELISA

SECONDARY OUTCOMES:
Changing IL-6 levels | 6 month
  Salivary and GCF level measured by ELISA
Changing IL-23 levels | 6 month
  Salivary and GCF level measured by ELISA
Changing IL-17E levels | 6 month
  Salivary and GCF level measured by ELISA